CLINICAL TRIAL: NCT00057044
Title: From Research to Practice - Lipid Management for Low HDL-Cholesterol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRX 01-083
Record Dates: First submitted 2003-03-27; First posted 2003-03-28 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Physicians' Practice Patterns; Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: education and reminder

INTERVENTIONS:
Behavioral: education and reminder

SUMMARY:
The overall purpose of this project is to improve the clinical outcomes of veterans with ischemic heart disease (IHD) through implementation of evidence-based lipid management, with a particular focus on veterans whose primary lipid abnormality is a low level of HDL-cholesterol (the �good� cholesterol).

DETAILED DESCRIPTION:
Background:

The overall purpose of this project is to improve the clinical outcomes of veterans with ischemic heart disease (IHD) through implementation of evidence-based lipid management, with a particular focus on veterans whose primary lipid abnormality is a low level of HDL-cholesterol (the �good� cholesterol).

Objectives:

The major objectives are 1. to determine whether a multifaceted intervention results in improved guideline-concordant lipid management for patients with low HDL-cholesterol; and 2. to test the relative effectiveness of three different reminder systems on physician prescribing behavior.

Methods:

The primary care clinic at each of the six VISN 13 facilities will serve as intervention sites. Within those sites we will randomize providers to one of three reminder systems. Control sites will consist of twelve other facilities matched to the intervention sites on the basis of facility characteristics. We will use a modified �pre-post� nested cohort design that allows us to evaluate the effect of the intervention controlling for secular trends. Target patients will be identified based on the following: 1. an IHD diagnosis within the past 5 years; 2. regular follow-up in a primary care clinic; 3. most recent LDL-cholesterol < 130 mg/dl and HDL-cholesterol < 40 mg/dl; 4. No lipid therapy within prior 6 months. The intervention will consist of: a. an on-site interactive educational workshop for providers; b. reminders (either patient-directed mailed reminders, computer-chart reminders at the time of visit, or automatic consults); c. opinion leader recruitment and �activation�. The primary outcome is proportion of target patients receiving guideline-concordant therapy. For objective 1, the outcome will be compared between intervention and control sites. For objective 2, the outcome will be compared between the three groups randomized to the different reminder systems. In addition, providers will be surveyed with a written questionnaire to determine their reaction to the educational workshop and the different reminder systems.

Status:

Intervention and data collection are completed. Data analysis is being undertaken, final report will soon follow.

ELIGIBILITY:
Inclusion Criteria:

Subjects are primary care providers from participating VISN sites. Patients whose medical records are utilized are selected via an algorithm.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11700 (Estimated)
Dates: Start 2001-10; Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hanna E. Bloomfield, MD MPH, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States